CLINICAL TRIAL: NCT05036798
Title: A Single-arm, Open, Phase II Clinical Study of Tislelizumab Combined With Lenvatinib and Gemox Regimen for Transformational Treatment of Potentially Resectable Locally Advanced Malignant Tumors of Biliary System.
Brief Title: Tislelizumab+Lenvatinib+Gemox Regiment for Potentially Resectable Locally Advanced Malignant Tumors of Biliary System.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDS20210220320615
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Potentially Resectable Locally Advanced Malignant Tumors of Biliary System
MeSH Terms: interventions — tislelizumab; lenvatinib; gemcitabine-oxaliplatin regimen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab combined with Lenvatinib and GEMOX (Experimental): Chemotherapy regimen(GEMOX):
  Gemcitabine 1g/m2,Oxaliplatin 100mg/m, D1, Q3W Tislelizumab 200mg D1 Q3w Lenvatinib 4mg Po QD
  Receive at least 3 cycles of combined treatment, and perform imaging evaluation after 3 cycles of treatment. If surgical treatment is not possible, imaging evaluation will be performed every two cycles thereafter until surgical treatment is feasible. If more than 7 cycles are still not possible for surgical resection, enter Tislelizumab + Lenvatinib maintenance treatment until the disease progresses or the toxicity cannot be tolerated.
  If patients undergoing R0 resection, start to receive Tislelizumab + Lenvatinib+Gemox regimen in 4-8 weeks after surgery for 7 cycles, and then entered Tislelizumab+Lenvatinib for 1 year or disease progression or toxicity cannot be tolerated
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Chemotherapy regimen:
  Gemcitabine 1g/m2 Oxaliplatin 100mg/m, D1, q3W2 Tislelizumab 200mg D1 Q3w Lenvatinib 4mg Po QD
  Other Names: Lenvatinib; Gemox

SUMMARY:
This is a single-arm, open, Phase II clinical study of Tislelizumab combined with lenvatinib and Gemox regimen for transformational treatment of potentially resectable locally advanced malignant tumors of biliary system.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histological diagnosis of potentially resectable local advanced biliary malignancies (intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, gallbladder carcinoma, ampullary carcinoma);

Potential resectable criteria: The first-stage R0 resection cannot be guaranteed for patients with cholangiocarcinoma admitted to our hospital, and there are the following imaging characteristics (satisfy one or more) :

1. The hilar and retroperitoneal lymph nodes were considered for metastasis but could be resected completely.
2. Intrahepatic cholangiocarcinoma has multiple foci, but foci are less than three and limited to half of the liver.
3. Local progression of gallbladder carcinoma with colon or duodenal involvement.
4. Hilar cholangiocarcinoma or lower segment of cholangiocarcinoma involving portal vein or hepatic artery requires combined vascular resection or reconstruction; 2. Patient age 20-79 years; 3. At least one measurable lesion as defined in RECIST version 1.1; 4. ECOG score was 0-1; 5. No prior medical treatment; 6. Adequate organ and bone marrow function and laboratory tests meet the following requirements:

   1. HGB≥90g/L；
   2. NEUT≥1.5×109/L；
   3. PLT ≥100×109/L；
   4. TBIL≤1.5 times normal upper limit (ULN);
   5. ALT and AST ≤2.5 x ULN;ALT and AST≤5×ULN for liver metastasis;
   6. Endogenous creatinine clearance ≥50ml/min (Cockcroft-Gault formula);
   7. Urinary protein < (++), or 24 hours urinary protein <1.0 g; 7. Coagulation was normal without active bleeding

   <!-- -->

   1. International standardized ratio INR≤1.5;
   2. Partial thrombin time APTT≤1.5 ULN; 8. Women of childbearing age must have a negative pregnancy test (serum or urine) within 14 days prior to enrollment and voluntarily use an appropriate method of contraception during the observation period and within 8 weeks after the last administration of the study drug;For men, surgical sterilization or consent to use appropriate methods of contraception during the observation period and for 8 weeks after the last administration of the study drug; 9. Estimated survival ≥3 months; 10. The patients voluntarily participated in the study and signed the informed consent (ICF); 11. It is expected that patients with good compliance will be able to follow up the efficacy and adverse reactions according to protocol requirements.

      12. Tumor tissue samples for PD-L1 expression analysis and microsatellite instability analysis.

      Exclusion Criteria:

      - The patient must be excluded from the study if any of the following conditions occur at the time of inclusion:

      1. Allergic to known anti-PD-1 and anti-PD-L1 antibodies; 2. Patients with hypertension (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg), grade I or above coronary heart disease, grade I arrhythmia (including prolonged QTc interval > 450 ms in males and > 470 ms in females) and grade I cardiac insufficiency; 3. Risk of biliary obstruction; 5. Allergic to the drugs of the program (gemcitabine, oxaliplatin); 6. Patients with a clear tendency of gastrointestinal bleeding, including the following conditions: local active ulcer lesions, and fecal occult blood (++) cannot be included in the group; Patients with a history of melena and hematemesis within 1 month; 7. Patients with immune system diseases need to take more than 10mg of dexamethasone daily; 8. Patients with concomitant diseases that, according to the judgment of the investigator, seriously endanger the patient's safety or affect the patient's ability to complete the study; 9. The researcher considered it unsuitable for inclusion.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 5 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 18 months
Disease control rate (DCR) | 5 months
Objective response rate (ORR) | 5 months
Overall survival (OS) | 24 months
Improvement in quality of life as measured by the EORTC Quality of Life Questionnaire QLQ-C30 (V3.0) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China